CLINICAL TRIAL: NCT05318534
Title: GL-0719 - A Phase 1, Double-blind, Placebo-controlled, Single Ascending Intravenous and Subcutaneous Injection Dose, Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Study in Healthy Male and Female Subjects and an Open-label Evaluation of Safety, Tolerability, Pharmacokinetics, and Pilot Efficacy Biomarkers in Subjects With Cold Agglutinin Disease
Brief Title: Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Study in Healthy Male and Female Subjects and Safety, Tolerability, Pharmacokinetics, and Pilot Efficacy Biomarkers in Subjects With Cold Agglutinin Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Gliknik Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: GL0719-01; 2021-004925-57 (EudraCT Number)
Record Dates: First submitted 2022-03-28; First posted 2022-04-08 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: First in Man Study to Evaluate Initial Safety
Keywords: complement-mediated diseases

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GL-0719 (Experimental): Dose level cohorts randomized in a 3:1 ratio to GL-0719 or placebo treatment, respectively.
  The study will comprise a single-dose, sequential-group design.
  Single Ascending IV Dose Cohorts
  * Cohort 1: 4 subjects
  * Cohort 2: 8 subjects
  * Cohort 3: 8 subjects
  * Cohort 4: 8 subjects
  * Cohort 5: 8 subjects
  Subcutaneous Injection Cohort
  * Cohort 6: 8 subjects
  * Cohort 7: 8 subjects
  * Cohort 8 (Patient Arm): Up to 6 subjects with Cold Agglutinin Disease (CAD); Placebo is not applicable.
  * Cohort 9 (Patient Arm): Up to 12 subjects with Cold Agglutinin Disease (CAD); Placebo is not applicable.
  Interventions: Drug: GL-0719
- Placebo (Placebo Comparator): Dose level cohorts randomized in a 3:1 ratio to GL-0719 or placebo treatment, respectively.
  The study will comprise a single-dose, sequential-group design.
  Single Ascending IV Dose Cohorts
  * Cohort 1: 4 subjects
  * Cohort 2: 8 subjects
  * Cohort 3: 8 subjects
  * Cohort 4: 8 subjects
  * Cohort 5: 8 subjects
  Subcutaneous Injection Cohort
  * Cohort 6: 8 subjects
  * Cohort 7: 8 subjects
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GL-0719 — Administration route: intravenous infusion and subcutaneous injection
  Arms: GL-0719
Drug: Placebo — Administration route: intravenous infusion and subcutaneous injection
  Arms: Placebo

SUMMARY:
The purpose of this first-in-human (FIH) study is to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of GL-0719 following single intravenous (IV) and subcutaneous injection (SC) doses in healthy adult male and female subjects.

In addition, safety, tolerability, PK, and pilot efficacy biomarkers will be evaluated in subjects with cold agglutinin disease (CAD).

ELIGIBILITY:
Inclusion Criteria for Cohorts 1 to 7

1. Healthy female or male subjects who, at the time of screening, are between the ages of 18 and 65 years, inclusive.
2. Females will not be pregnant or lactating, and females of childbearing potential and males will agree to use contraception.
3. Body mass index of 18.0 to 32.0 kg/m^2, inclusive; and a total body weight > 50 kg up to a maximum of 110 kg.
4. Study subjects must have received a quadrivalent meningococcal conjugate vaccine (meningococcal serogroups A, C, W, and Y) within the past 5 years or vaccination a minimum of 14 days prior to initial study drug administration.
5. The subject must be capable of understanding the investigational nature, potential risks and benefits of the study and capable of providing valid informed consent.

Inclusion Criteria for Cohorts 8 to 9

1. Female or male subjects who, at the time of screening, are at least 18 years of age with a total body weight of ≥ 50 kg.
2. Females will not be pregnant or lactating, and females of childbearing potential and males will agree to use contraception.
3. The subject must be capable of understanding the investigational nature, potential risks and benefits of the study and capable of providing valid informed consent.
4. The subject must be willing to return to the study center for study treatment and study-related follow-up procedures as required by the protocol.
5. Study subjects must have received a quadrivalent meningococcal conjugate vaccine (meningococcal serogroups A, C, W, and Y) within the past 5 years or vaccination a minimum of 14 days prior to initial study drug administration.
6. The Participant Identification Center (PIC) site will have provided evidence that the PIC site used to confirm diagnosis of Cold Agglutinin Disease (CAD)
7. Primary Cold Agglutinin Disease (CAD) or CAD secondary to active lymphoid or other hematologic malignancy (Cold Agglutinin Syndrome).
8. Hemoglobin level < 105 gram per liter (g/L).
9. Bilirubin level above the normal reference range.

Key Exclusion Criteria for Cohorts 1 to 7

1. History of any clinically significant (as determined by the investigator) cardiac, endocrine, hematological, hepatic, immunological, metabolic, urological, pulmonary, neurological, dermatological, psychiatric, renal, or other major disease.
2. Evidence of clinically significant medical condition or other condition that might significantly interfere with the absorption, distribution, metabolism, or excretion of study drug, or place the subject at an unacceptable risk as a participant in this study.
3. Signs and symptoms of, or diagnosis consistent with a chronic autoimmune disorder and/or positive antinuclear antibodies (ANA) test by indirect immunofluorescence confirmed by ANA titer ≥ 1:160.
4. Documented history of autoimmune disease, or history of a syndrome that required systemic steroids or immunosuppressive medications, except for subjects with vitiligo or resolved childhood asthma/atopy.
5. Any underlying medical condition that, in the opinion of the investigator, renders the subject a poor candidate for this study or could confound the results of the study or put the subject at undue risk.

Key Exclusion Criteria for Cohorts 8 to 9

1. CAD secondary to infection or an autoimmune disorder.
2. CAD secondary to active lymphoid or other hematologic malignancy not meeting the inclusion criteria.
3. Diagnosis of any other malignancy except for adequately treated basal or squamous cell skin cancer, curatively treated in situ disease, or other cancer from which the subject has been disease-free for ≥ 5 years.
4. Clinically relevant infection of any kind within the month preceding enrollment (example, active hepatitis C, pneumonia).
5. Clinical diagnosis of Systemic Lupus Erythematosus (SLE), other autoimmune disorders, or ANA titer > 1:160 at Screening.
6. Positive hepatitis panel and/or positive HIV (Human Immuno Deficiency) test. Subjects whose results are compatible with prior immunization may be included at the discretion of the investigator.
7. Positive HIV antibody at Screening.
8. Treatment with an investigational drug within 90 days or five half-lives preceding the first dose of IP (whichever is longer), with the exception of subjects who received GL-0719 in this study in Cohort 8, who cannot be re-enrolled in Cohort 9 within 60 days after their last dose of GL-0719.
9. Concurrent plasma exchange therapy.

Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-04-08 (Actual); Primary Completion 2026-01-21 (Estimated); Study Completion 2026-01-21 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) | Day 1 to Follow-up (Day 31±2)
Incidence of laboratory abnormalities, based on hematology, clinical chemistry, and urinalysis test results | Screening (Days -42 to -15) to Follow-up (Day 31±2)
Incidence of abnormal clinical laboratory findings in 12-lead ECG parameters, vital signs, physical examination and measurement of cytokines | Screening (Days -42 to -15) to Follow-up (Day 31±2)

SECONDARY OUTCOMES:
Area Under the Concentration time Curve from Time 0 Extrapolated to Infinity (AUC0-∞) | Day 1 to Follow-up (Day 31±2)
Area Under the Concentration time Curve from Time 0 to the Time of the Last (AUC0-tlast) | Day 1 to Follow-up (Day 31±2)
Maximum Observed Concentration (Cmax) | Day 1 to Follow-up (Day 31±2)
Time of the maximum observed concentration (tmax) | Day 1 to Follow-up (Day 31±2)
Apparent terminal elimination half-life (t1/2) | Day 1 to Follow-up (Day 31±2)
For Cohorts 1 to 7: The degree of complement classical pathway inhibition in study subjects over time as evaluated by the MicroVue CH50 Eq EIA assay | Day 1 to Follow-up (Day 31±2)
Incidence of anti-drug antibodies | Day -1, Day 15±1 and Follow-up (Day 31±2)

CONTACTS AND LOCATIONS:
Overall Officials: Jim Bush, MBChB, PhD, Principal Investigator — Fortrea Clinical Research Unit Ltd.
Locations (1):
- Fortrea Clinical Research Unit Ltd, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No